CLINICAL TRIAL: NCT03254589
Title: Methotrexate, Blood Pressure and Arterial Function in Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Flinders University (Other)
Collaborators: University of South Australia (Other); medac GmbH (Industry)
Responsible Party: Principal Investigator, Arduino Mangoni, Professor of Clinical Pharmacology, Flinders University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HREC/17/SAC/46
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Rheumatoid Arthritis; Stiffness, Aortic; Endothelial Dysfunction; Cardiovascular Risk Factor
Keywords: Methotrexate; Rheumatoid arthritis; Blood pressure; Arterial stiffness; Cardiovascular risk
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Sulfasalazine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Experimental): Newly diagnosed RA patients started on subcutaneous MTX - open randomisation vs. sulfasalazine. In this group, use of NSAIDs, steroids, and/or other DMARDs, is allowed, if indicated, for symptom control. The overall management, tests and outpatient rheumatology visits schedule will be similar to other patients with RA, in accordance to standard practice .
  Interventions: Drug: Methotrexate
- Group 2 (Active Comparator): Newly diagnosed RA patients started on sulfasalazine - open randomisation vs. subcutaneous MTX. In this group, use of NSAIDs, steroids, and/or other DMARDs (except MTX), is allowed, if indicated, for symptom control. The overall management, tests and outpatient rheumatology visits schedule will be similar to other patients with RA, in accordance to standard practice.
  Interventions: Drug: Sulfasalazine
- Group 3 (Experimental): RA patients on long-term treatment (> 1 year) with oral MTX, with or without other DMARDs, NSAIDs and/or steroids, switched to subcutaneous MTX (same dose). In these patients, treatment with other DMARDs, NSAIDs and/or steroids will continue. The overall management, tests and outpatient rheumatology visits schedule will be similar to other patients with RA, in accordance to standard practice.
  Interventions: Drug: Methotrexate
- Group 4 (Active Comparator): RA patients on stable treatment (> 1 year) with other (non-MTX) DMARDs, with or without NSAIDs and/or steroids, and continued on the same treatment. The overall management, tests and outpatient rheumatology visits schedule will be similar to other patients with RA, in accordance to standard practice.
  Interventions: Drug: Other DMARDs

INTERVENTIONS:
Drug: Methotrexate — See arm descriptions
  Arms: Group 1; Group 3
Drug: Sulfasalazine — See arm description
  Arms: Group 2
Drug: Other DMARDs — See arm
  Arms: Group 4

SUMMARY:
The investigators will study the effects of methotrexate on blood pressure, arterial stiffness and endothelial function in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Patients with rheumatoid arthritis have an increased risk of stroke and heart attack when compared to the rest of the population. Recent studies have shown that methotrexate, a disease-modifying antirheumatic drug (DMARDs) commonly prescribed for rheumatoid arthritis, reduces this risk. However, the mechanisms responsible for the protective effects of methotrexate on the heart and the brain are unknown.

The investigators have recently completed an observational study in participants with rheumatoid arthritis treated with either methotrexate or with other DMARDs. Participants on methotrexate had lower blood pressure and 'healthier' blood vessels than participants treated with other DMARDs. These differences were maintained over a period of 8 months. These results suggest that methotrexate lowers blood pressure and exerts salutary effects on blood vessels, which might explain the reduced risk of stroke and heart attack with this drug. However, the observational nature of this study does not allow establishing a clear cause-effect relationship between methotrexate treatment and the observed changes in blood pressure and blood vessels.

In order to address this issue, the investigators will recruit participants that have been recently diagnosed with rheumatoid arthritis and are about to start treatment with either methotrexate (Group 1) or another DMARD (Group 2). Then, the investigators will assess their blood pressure and blood vessels for 6 months. The investigators will use an injectable (subcutaneous) form of methotrexate because this might provide better effects on blood pressure and blood vessels. The investigators will also study a third group (Group 3) of rheumatoid arthritis participants already on treatment (> 1 year) with oral methotrexate, with or without other DMARDs. They will be switched to subcutaneous methotrexate, but continuing all their other medications, for 6 months to see whether the subcutaneous form can further reduce blood pressure and provide additional salutary effects on blood vessels. Finally, the investigators will study a fourth group (Group 4) of participants with rheumatoid arthritis already on treatment (> 1 year) with DMADRs other than methotrexate who will continue with the same medications for 6 months, to assess possible fluctuations in blood pressure and blood vessel markers over time.

Each participant will attend three study visits (baseline, 1 and 6 months), each lasting between 60 and 90 min.

ELIGIBILITY:
Inclusion Criteria:

* Patient with rheumatoid arthritis according to EULAR/ACR 2010 criteria.
* Age ≥18 years.
* Written informed consent, dated and signed before initiating any study-related procedure.

Exclusion Criteria:

* Contraindication to MTX or sulfasalazine.
* Patient who cannot be followed during 6 months.
* Active alcohol or substance abuse within the last 12 months.
* Participation in a clinical trial within 3 months prior to the start of the study.
* Body mass index >35 Kg/m2.
* Secondary causes of hypertension.
* Grade 2 (moderate) or 3 (severe) hypertension: clinic blood pressure >160/100 mm Hg.
* Resistant hypertension: clinical blood pressure ≥140/90 mm Hg despite concurrent use of three antihypertensive agents of different classes, one of which is a diuretic.
* Clinical systolic blood pressure <100 mm Hg or history of symptomatic orthostatic hypotension.
* Cardiovascular event, procedure, or hospitalization for unstable angina with the last 6 months.
* Atrial fibrillation.
* Heart failure.
* Treatment with nitrates.
* Estimated glomerular filtration rate (eGFR) <45 mL/min.
* Diagnosis of polycystic kidney disease.
* Glomerulonephritis treated with or likely to be treated with immunosuppressant drugs
* Uncontrolled diabetes with HbA1c >9.0% (>75 mmol/mol).
* Uncontrolled dyslipidaemia with total serum cholesterol >7.5 mmol/L or triglycerides >5.6 mmol/L.
* Clinical diagnosis of dementia, treatment with medications for dementia or, in the opinion of the study staff, the participant is cognitively unable to follow the protocol.
* Other medical, psychiatric, or behavioural factors that in the judgment of the study staff may interfere with study participation.
* Cancer diagnosed and treated within the past 2 years that, in the judgment of the study staff, would compromise a participant's ability to comply with the protocol and complete the study.
* Any organ transplant.
* Pregnancy, currently trying to become pregnant, or of child bearing potential and not using birth control.
* Significant illness within 2 weeks of study start.
* Patients with an unstable active medical condition that could impair evaluation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in peripheral systolic blood pressure | Change from baseline peripheral systolic blood pressure at 6 months
  Change in peripheral systolic blood pressure

SECONDARY OUTCOMES:
Change in peripheral and central blood pressure | Change from baseline peripheral and central blood pressure at 6 months
  Change in peripheral and central blood pressure
Change in arterial stiffness | Change from baseline pulse wave velocity at 6 months
  Change in pulse wave velocity
Change in arterial wave reflection | Change from baseline augmentation index at 6 months
  Change in augmentation index
Change in adenosine | Change from baseline adenosine concentrations at 6 months
  Change in adenosine concentrations
Change in arginine metabolites | Change from baseline ADMA concentrations at 6 months
  Change in ADMA concentrations

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Adelaide Local Health Network, Bedford Park, South Australia, Australia

REFERENCES:
- [Derived] Mangoni AA, Wiese MD, Woodman RJ, Sotgia S, Zinellu A, Carru C, Hulin JA, Shanahan EM, Tommasi S. A controlled comparative study of the effects of methotrexate and pharmacogenetic factors on arterial blood pressure and arterial stiffness in patients with rheumatoid arthritis. Ann Med. 2025 Dec;57(1):2539311. doi: 10.1080/07853890.2025.2539311. Epub 2025 Jul 31. PMID 40742006
- [Derived] Mangoni AA, Wiese MD, Woodman RJ, Sotgia S, Zinellu A, Carru C, Hulin JA, Shanahan EM, Tommasi S. Methotrexate, blood pressure and arterial function in rheumatoid arthritis: study protocol. Future Cardiol. 2024;20(13):671-683. doi: 10.1080/14796678.2024.2411167. Epub 2024 Oct 10. PMID 39387403

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT03254589/Prot_SAP_000.pdf